CLINICAL TRIAL: NCT07384819
Title: Evaluation of Visual Perception Development in Autism: Duration of a Moment
Brief Title: Duration of Moment in Autism
Acronym: DOMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A02488-41
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; Prototypical autism; Temporal Integration Window; Attentional Blink; Eye-tracking; Visual perception; Infant development
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Neurotypical 3-year-olds (Other): 3-year-old children without a neurodevelopmental disorder
  Interventions: Behavioral: Temporal Integration Window task; Behavioral: Attentional Blink task
- Neurotypical 5-year-olds (Other): 5-year-old children without a neurodevelopmental disorder
  Interventions: Behavioral: Temporal Integration Window task; Behavioral: Attentional Blink task
- Prototypical ASD 3-year-olds (Experimental): 3-year-old children with a diagnosis of ASD and prototypical characteristics
  Interventions: Behavioral: Temporal Integration Window task; Behavioral: Attentional Blink task
- Prototypical ASD 5-year-olds (Experimental): 5-year-old children with a diagnosis of ASD and prototypical characteristics
  Interventions: Behavioral: Temporal Integration Window task; Behavioral: Attentional Blink task
- Non-prototypical ASD 3-year-olds (Experimental): 3-year-old children with a diagnosis of ASD but not prototypical characteristics
  Interventions: Behavioral: Temporal Integration Window task; Behavioral: Attentional Blink task
- Non-prototypical ASD 5-year-olds (Experimental): 5-year-old children with a diagnosis of ASD but not prototypical characteristics
  Interventions: Behavioral: Temporal Integration Window task; Behavioral: Attentional Blink task

INTERVENTIONS:
Behavioral: Temporal Integration Window task — The TIW task involves alternating visual displays (integration and segmentation trials) across four inter-stimulus intervals (ISI: 16, 32, 83, 116 ms). This task allows estimation of the participant's perceptual integration threshold.
Behavioral: Attentional Blink task — The Attentional Blink task presents rapid sequences of images (including two targets and distractors), measuring the minimum time delay required for both targets to be detected. Three different T1-T2 intervals are tested.

SUMMARY:
This study investigates the temporal dynamics of perception and attention in children with Autism Spectrum Disorder (ASD), focusing on two key phenomena: the Temporal Integration Window (TIW) and the attentional blink. Using eye-tracking, 3- and 5-year-old children with ASD (prototypical or not) will be compared to age-matched neurotypical peers.

The investigators hypothesize that children with ASD exhibit shorter TIWs and attentional blinks, reflecting faster perceptual sampling and attentional processing. These characteristics may contribute to sensory hypersensitivity and difficulties in complex, unpredictable environments such as social situations. The protocol includes two experimental tasks.

DETAILED DESCRIPTION:
The study is a multicenter research project that aims to investigate the temporal dynamics of visual perception and attention in children with Autism Spectrum Disorder (ASD), including both prototypical and non-prototypical subgroups. It compares these groups to age-matched neurotypical peers. The study focuses on two distinct cognitive phenomena:

Temporal Integration Window (TIW) : a pre-attentive perceptual mechanism that determines the time frame within which visual information is integrated into a unified percept. In typically developing adults, this window is estimated to be around 65 milliseconds. Prior research suggests that children with ASD may have a shorter TIW, indicating faster perceptual sampling.

Attentional Blink (AB) : a post-perceptual phenomenon reflecting limitations in attentional resources. When two targets are presented in rapid succession, the second target is often missed if it follows too closely after the first. The duration of the attentional blink is thought to decrease with age and maturation. Previous studies have shown that attentional blink is already present at 5 months of age and shortens during development.

The central hypothesis is that both TIW and AB durations might be shorter in children with ASD, reflecting faster perceptual and attentional processing. This accelerated dynamic could contribute to sensory hypersensitivity and difficulty coping with complex or unpredictable environments, such as those involving social stimuli.

A total of 228 children will participate, divided into six groups.

Each participant will complete two eye-tracking tasks during a single session lasting approximately one hour:

* The TIW task
* The Attentional Blink task

Developmental level is assessed using validated tools: the Mullen Scales of Early Learning, VINELAND-2 or the IDE questionnaire, depending on the child's group.

The study will also examine whether the prototypical ASD subgroup, as defined by clinical criteria shows distinct perceptual profiles, and whether age or developmental level influences temporal dynamics.

This study aims to better understand early perceptual and attentional processes in autism.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 or 5 years
* Either with a diagnosis of Autism Spectrum Disorder (ASD) or typically developing (neurotypical)
* No intellectual disability (per Mullen, Denver, or psychometric report)
* Normal or corrected vision and hearing
* Written informed consent from legal guardians
* Legal guardians affiliated to a French social security plan
* For ASD group only : classification as prototypical or non-prototypical based on clinical evaluation

Exclusion Criteria:

* Neurological disorder
* Parental or child refusal to participate
* For neurotypical children: developmental delay or psychiatric diagnosis

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 228 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-08-16 (Estimated); Study Completion 2028-08-16 (Estimated)

PRIMARY OUTCOMES:
Temporal dynamics of perception | Baseline
  The Temporal Integration Window (TIW) is defined as the shortest interval between two displays that can be integrated into a single percept
Temporal dynamics of attention | Baseline
  The Attentional Blink duration, defined as the minimal delay between two target stimuli that allows detection of both.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Baby lab - Institut des sciences cognitives Marc Jeannerod, Bron
  - CEDA - Le Vinatier, Bron

IPD SHARING:
Plan to Share IPD: Yes